CLINICAL TRIAL: NCT03020576
Title: Robot-assisted Hand Training (Amadeo) Compared With Conventional Physiotherapy Techniques in Chronic Ischemic Stroke Patients: A Pilot Study
Brief Title: Robotic and Conventional Hand Therapy After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Medical University Innsbruck (Other); New York University (Other)
Responsible Party: Principal Investigator, Joel Stein, Department of Rehabilitation and Regenerative Medicine Chair, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAI0093
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Therapy (Active Comparator): Participants randomized to this arm will receive conventional based therapy to their affected upper limb dose matched with the Robotic Therapy group. These interventions are aimed at increasing range of motion, strength and function at the shoulder, elbow, wrist and hand.
  Interventions: Other: Conventional Therapy
- Robotic Therapy (Experimental): Participants randomized to this arm will receive robotic based therapy using the Amadeo Hand Robot device to improve range of motion, strength, and coordination to the wrist and hand.
  Interventions: Device: Amadeo Hand Robot Device

INTERVENTIONS:
Device: Amadeo Hand Robot Device — This is a robotic device designed to offer rehabilitation to remediate weakness and limitations of range of motion of the hand and fingers.
  Arms: Robotic Therapy
Other: Conventional Therapy — This arm involves treatment using conventional methods designed to promote range of motion, strength, coordination and function at the level of the shoulder, elbow, wrist and hand.
  Arms: Conventional Therapy

SUMMARY:
Weakness is a major cause of disability in stroke survivors. Rehabilitation techniques are often not effective in restoring full function of the upper limb. Specifically, many individuals remain with weakness in the hand, preventing its return to full use.

Robotic therapies have been developed as exercise tools for stroke survivors. Devices, such as the InMotion2, have been shown to be useful in restoring some motor function in the upper limb. However, most existing devices designed to be used with the upper limb have primarily been developed to treat the shoulder, elbow and wrist. They have not specifically addressed hand function.

Tyromotion, Inc. has developed the Amadeo, which is primarily intended to provide rehabilitation for patients with neurological or orthopedic deficits in hand function. Initial clinical testing has demonstrated the practicality of using this device in a population of stroke survivors, although further research is needed to better understand the usefulness of the Amadeo device as compared with conventional rehabilitation methods. The purpose of this study was to compare results of training with the Amadeo device or training with conventional therapies.

A total of 28 subjects from two separate sites participated in the study and underwent baseline testing of upper limb motor and sensory performance and function. Subjects were then assigned to one of two treatment groups with a 50:50 chance of being in either group. One group underwent training with the Amadeo device and the other group underwent training with conventional therapy. All training sessions were 60 minutes in duration, three days/week for eight weeks (24 total sessions). Subjects were reassessed on completion of the training program.

ELIGIBILITY:
Inclusion Criteria:

* history of stroke (>3 months from time of ictus)
* paresis or plegia of the upper extremity.

Exclusion Criteria:

* severe spasticity (defined on the Ashworth Scale with a score of 4-5)
* severe pain despite conventional pain therapy of the paretic upper extremity
* swelling, infection, fracture or ulcers of the paretic extremity
* arthritis of the hand joints
* pregnant
* botulinum toxin- therapy to the upper extremity within 3 months prior to study entry
* severe contractions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stein, MD, Principal Investigator — Columbia University; Raimund Helbok, MD, Principal Investigator — Innsbruck Medical University
Locations (2):
- Columbia University Medical Center, New York, New York, United States
- Innsbruck Medical University, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Group: The purpose of this group is to provide training that is matched to the robotic group in duration and intensity. Participants randomized to this group receive therapy to the affected/paretic upper limb. This therapy is aimed at improving range of motion, strength and functionality. Similar to the robotic group, treatment sessions occurred three times weekly for eight weeks, and sessions were 60 minutes in duration.
- Robotic Group: The purpose of this group was to provide robotic based training using the Amadeo Hand Robotic Device (Tyromotion, GmbH, Graz, Austria) as a tool to improve range of motion, strength and functionality of the hand in a population of individuals post stroke. Treatment sessions were conducted three times weekly over eight weeks. Each session was 60 minutes in duration.
Period: Overall Study
Arm/Group | Conventional Group | Robotic Group
Started | 15 | 16
Completed | 14 | 14
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Group | Robotic Group | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.14 (17.9) | 54.57 (13.8) | 57.13 (15.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 11 | 7 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 10 | 6 | 16
  United States | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Impairment Based Arm Measures - Change in Upper Extremity Portion of the Fugl Meyer
Description: quantitative performance measure (scale ranging from 0 (minimum) to 66 (maximum) points) of arm and hand impairment. A higher score represents more skilled movements of the arm and hand.
Time Frame: Through study completion, an average of 8 weeks (at baseline and at the 8-week completion point)
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Conventional Group | Robotic Group
Number analyzed (Participants) | 14 | 14
change in units on a scale | 5.9 (13.7) | 2.1 (16.3)

2. Secondary Outcome: Change in Range of Motion Measures
Description: quantitative assessment of the mobility of joints throughout the upper limb using standard goniometric measures. Measured in degrees (0-360 degrees)
Time Frame: Through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Conventional Group | Robotic Group
Number analyzed (Participants) | 14 | 14
change in units on a scale | 3.53 (0.45) | 3.33 (0.80)

3. Secondary Outcome: Change in Hand and Pinch Strength
Description: quantitative assessment of hand strength using standard dynamometry measurements in units of kilograms
Time Frame: Through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: change in kilograms
Arm/Group | Conventional Group | Robotic Group
Number analyzed (Participants) | 14 | 14
change in kilograms | 1.63 (7.8) | 0.84 (5.3)

4. Secondary Outcome: Change in Motor Activity Log Amount
Description: quantitative, self report scale measuring the 'Amount' and 'How Well' an individual performs a battery of motor tasks. Maximum score of 150 (raw score) for each 'Amount' and 'How Well' sections. Higher scores reflect better performance.
Time Frame: Through study completion (taken at baseline and at 8-week study completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Group | Robotic Group
Number analyzed (Participants) | 14 | 14
units on a scale | 9.35 (35.1) | 2.53 (37.7)

5. Secondary Outcome: Change in Mobility and Activities of Daily Living
Description: The Barthel Index is a quantitative scale measuring the need for assistance an individual has in performance of tasks of general mobility and activities of daily living. Maximum raw score is 100. Higher values represent better outcomes.
Time Frame: Through study completion (taken at baseline and at 8 week study completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Group | Robotic Group
Number analyzed (Participants) | 14 | 14
units on a scale | 6.78 (19.1) | -0.36 (12.3)

6. Secondary Outcome: Change in Hand Dexterity
Description: The 9 Hole Peg Test was used as a quantitative measure of hand dexterity. The participant is asked to remove the pegs and put them back into the slots in a period of 100 sec. The number of pegs moved is recorded as an overall score.
Time Frame: Through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Group | Robotic Group
Number analyzed (Participants) | 14 | 14
units on a scale | 10.67 (47.8) | -1.12 (24.3)

7. Secondary Outcome: Change in Spasticity Measures
Description: The Modified Ashworth Scale is a standardized quantitative assessment of muscle tightness/spasticity during movements of the arm and wrist. It is scored on a scale of 1-5, with higher numbers reflecting a greater severity of spasticity.
Time Frame: Through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Conventional Group | Robotic Group
Number analyzed (Participants) | 14 | 14
change in units on a scale | -0.10 (0.3) | -0.10 (0.2)

8. Secondary Outcome: Change in Motor Activity Log How Well
Description: as for outcome 4
Time Frame: Through study completion (taken at baseline and on 8 week study completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Group | Robotic Group
Number analyzed (Participants) | 14 | 14
units on a scale | 12.79 (29.5) | 2.6 (35.4)

ADVERSE EVENTS:
Arm/Group | Conventional Group | Robotic Group
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No